CLINICAL TRIAL: NCT03412331
Title: Clinical And Microbiological Evaluations Of Adjunctive Photodynamic Therapy To Non-Surgical Periodontal Treatment In Patients With Generalized Aggressive Periodontitis
Brief Title: Effects Of Adjunctive Photodynamic Therapy To Non-Surgical Periodontal Treatment In Patients With Generalized Aggressive Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Borekci et al.
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Generalized Aggressive Periodontitis
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (2):
- Control Group (Active Comparator): NPT including scaling and root planing was applied to 12 subjects with ultrasonic and hand instruments until the operator feels that root surface is clean, hard and smooth.
  Interventions: Device: Ultrasonic; Device: Hand Instruments
- Test Group (Experimental): Following NPT, toluidine blue O mediated PDT was performed with a LED source (625-635 nm wavelength) (FotoSan®, CMS Dental, Denmark) to 12 subjects. The dye (0.1 mg/ml) was applied with a canula into the periodontal pockets. After 3 minutes, the subjects rinsed their mouths with sterile saline solution for removal of excessive dye. Then, the applicator of photosensitizer was inserted until the bottom of the periodontal pocket and photoinactivation was performed in 6 sites per tooth for 10 seconds of each sites with a total of 60 seconds per tooth.
  Interventions: Device: Ultrasonic; Device: Hand Instruments; Device: LED Source

INTERVENTIONS:
Device: Ultrasonic — Cavitron® BOBCAT® Pro, Dentsply International, USA
Device: Hand Instruments — Gracey, SG 5/6, 7/8, 11/12, 13/14, Hu-Friedy Ins. Co., USA
Device: LED Source — LED source (625-635 nm wavelength) (FotoSan®, CMS Dental, Denmark)
  Arms: Test Group

SUMMARY:
Generalized aggressive periodontitis (GAgP) is a distinct type of periodontal disease characterized by rapid loss of attachment and alveolar bone occuring in young individuals. Photodynamic therapy (PDT) was introduced in periodontology as an adjunctive approach to non-surgical periodontal treatment (NPT) in periodontitis patients. In this trial, it was aimed that to evaluate the clinical and microbiological effects of adjunctive PDT to NPT in patients with GAgP. In this prospective controlled clinical study, 24 systemically healthy, non-smoking subjects with GAgP were enrolled. Subjects were randomly assigned to a control group (n=12) treated with NPT only or to a test group (n=12) treated with NPT and PDT. Plaque index, sulcus bleeding index (SBI), pocket depth (PD), relative attachment level, gingival recession, mobility were recorded at baseline and on day 63. Microbiological samples were obtained fom the sites with PD ≥5 mm at the same time points and evaluated for Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia and Treponema denticola using micro-IDent test.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy,
* non-smoker
* not received any periodontal treatment within the last 6 months
* no antibiotics, anti-inflammatory drugs or any other medication taken within the last 6 months
* consent to participate in the study

Exclusion Criteria:

* any systemic disease (i.e. diabetes mellitus, HIV infection) that might influence the prognosis of periodontal disease and outcome of the treatment
* any medical condition that required antibiotic prophylaxis before the treatment
* smoking
* pregnancy and lactation
* ingestion of antibiotics, anti-inflammatory drugs or any other medication during study period
* any physical limitations or restrictions that might preclude normal oral hygiene procedures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Probing Depth | 63 day
  defined as the distance from the free gingival margin to the bottom of the periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: Leyla KURU, Prof. Dr., Study Director — Marmara University, Faculty of Dentistry, Department of Periodontology

IPD SHARING:
Plan to Share IPD: No